CLINICAL TRIAL: NCT00749060
Title: Prospective Randomized Comparative Study of Balloon Kyphoplasty,Vertebroplasty and Conservative Management in Acute Osteoporotic Vertebral Fractures of Less Than 6 Weeks
Brief Title: Comparison of Balloon Kyphoplasty, Vertebroplasty and Conservative Management in Acute Osteoporotic Vertebral Fractures
Acronym: OSTEO-6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P060107
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Osteoporotic Vertebral Fracture; Between T5 and L5; of Less Than 6 Weeks Duration
Keywords: osteoporosis; non-traumatic vertebral fracture; vertebral compression; Balloon kyphoplasty; vertebroplasty
MeSH Terms: conditions — Osteoporosis | interventions — Kyphoplasty; Vertebroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Other): conventional treatment
  Interventions: Other: conventional treatment
- 2 (Other): kyphoplasty by balloons
  Interventions: Procedure: kyphoplasty with balloons
- 3 (Other): vertebroplasty
  Interventions: Procedure: vertebroplasty

INTERVENTIONS:
Other: conventional treatment — with our without brace
  Other Names: antalgic drugs
  Arms: 1
Procedure: kyphoplasty with balloons — Balloon Kyphoplasty which consists of placing through a percutaneous posterior approach under radiological guidance, into the fractured vertebra a balloon which is inflated with fluid and creates a cavity. This may restore part of the vertebral height loss due to the fracture. In addition, after balloon deflation, polymethylmetacrylate cement is injected with low pressure into the created cavity.
  Arms: 2
Procedure: vertebroplasty — Vertebroplasty consisting in the percutaneous injection into the fractured vertebra of polymethylmetacrylate cement (the cement used to fix prosthesis in joint replacement) through a posterior route through the vertebral pedicles under radiological guidance
  Arms: 3

SUMMARY:
This study aims to compare three treatments in recent (less than 6 week duration) non-traumatic ( usually osteoporotic) vertebral fractures.

DETAILED DESCRIPTION:
The three treatments are the following: 1/Conventional medical treatment including rest and pain medications2/Vertebroplasty consisting in the percutaneous injection into the fractured vertebra of polymethylmetacrylate cement (the cement used to fix prosthesis in joint replacement) through a posterior route through the vertebral pedicles under radiological guidance.3/Balloon Kyphoplasty which consists of placing through a percutaneous posterior approach under radiological guidance, into the fractured vertebra a balloon which is inflated with fluid and creates a cavity. This may restore part of the vertebral height loss due to the fracture. In addition, after balloon deflation, polymethylmetacrylate cement may be injected with low pressure into the created cavity. The study will indicate if balloon kyphoplasty is able to restore vertebral height of the fractured vertebra better than medical treatment and vertebroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to undergo the vertebroplasty or Balloon kyphoplasty procedure
* Patient must have signed the consent form (ZELEN Randomization protocol)
* Male or female, 50 years or older
* One or two non-traumatic vertebral fracture(s):

  * Of osteoporotic origin (low speed trauma such as fall from his own height or less than 80 cm)
  * Fracture(s) of less than 6 weeks duration after the onset of pain related to the fracture The fracture(s) exhibit(s) high signal intensity on T2-weighted images and a benign appearance at MRI
* The patient will be able to receive the selected protocol treatment within 6 weeks after onset of fracture-related symptoms and within 15 days after treatment randomization.
* The benign nature of the vertebral fracture has to be confirmed by the results of the biopsy performed during vertebroplasty or balloon kyphoplasty or by one year follow-up in the conservative treatment group.

Exclusion Criteria:

* Patient with a vertebral fracture of more than 6 week duration after onset of fracture-related symptoms.
* Neurological signs related to the vertebral fracture to treat
* History of surgical or percutaneous spine treatment except simple discectomy at a single or multiple vertebral levels with no residual pain.
* More than two recent vertebral fractures
* Current infection
* Impossibility to perform the percutaneous approach of the vertebra to treat.
* Reduction by more than 50% of the anteroposterior width of the bony spinal canal due to the vertebral fracture to treat.
* Known allergy to a contrast media or to one of the cement components used for kyphoplasty.
* Vertebral fracture with loss of 90%or more of the vertebral body height
* Neurological signs or symptoms related to the vertebral fracture
* Malignant and traumatic vertebral fractures
* Contraindication to MRI :

  * Metallic implant : pace-maker, non movable auditive implant, metallic vascular or cardiac device
  * Metallic surgical clips
  * Claustrophobia
* Evolutive cardiac disease nonreactive to medical treatment
* Patient presenting a non correctable spontaneous or therapeutic coagulation disorder.
* Presence of an unexplained biological inflammatory syndrome with NFS≥20
* Non compliant patient: Impossibility to participate to the study and to be followed up for 1 year.
* Pregnant or breast feeding women
* Patient not affiliated to social security

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in Vertebral Kyphotic angle between preoperative and one-year follow-up measurements. | 1 year

SECONDARY OUTCOMES:
1° - Pain evaluation using a visual analogic scale | J-20 à J-7 / J6 / J45 /J90 /J180 / J360
questionnaire (Eifel) for back pain evaluation | J-20 à J-7 / J6 / J45 /J90 /J180 / J360
Quality of life evaluation (QUALEFFO - Short-Form SF12). | J-20 à J-7 / J6 / J45 /J90 /J180 / J360
Analgesics intake according to the WHO classification (Classes 1, 2 and 3). | J-20 à J-7 / J6 / J45 /J90 /J180 / J360
Regional spine Kyphosis angle and global thoracic and lumbar Kyphosis angle | J-20 à J-7 / J6 / J45 /J90 /J180 / J360
Changes in anterior, mid and posterior vertebral heights of the treated vertebral body | J-20 à J-7 / J6 / J45 /J90 /J180 / J360
Changes in height of the intervertebral disc spaces adjacent to the treated vertebra | J-20 à J-7 / J6 / J45 /J90 /J180 / J360
Number of new vertebral fractures occurring during the one year follow-up period | J-20 à J-7 / J6 / J45 /J90 /J180 / J360
Cost evaluation in a sample of 10% of patients randomly selected including the following costs : o Intervention cost. o Medical treatment costs o Consultation costs. o Hospitalization cost o Complication costs | J-20 à J-7 / J6 / J45 /J90 /J180 / J360
Follow-up of anterior, median and posterior height of the treated vertebral body, obtained by making an average of all measurements, on 3 cuts tomodensitometry (tdm) on the sagittal level : lateral right, median and lateral left | preoperative, at J6 and at J360
Intensity of signal with T2 sequence | preoperative and at J360

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Denis LAREDO, MD,Pr, Principal Investigator — AP-HP Assistance Publique- Hôpitaux de Paris
Locations (1):
- Hopital LARIBOISIERE Service de Radiologie Ostéo-Articulaire, Paris, France